CLINICAL TRIAL: NCT06702956
Title: Assessment of Dimensional Bony Changes Following Laser Corticotomy in Rapid Canine Retraction
Brief Title: Assessment of Dimensional Bony Changes Following Laser Corticotomy
Acronym: Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Assessment of bony changes
Record Dates: First submitted 2024-11-03; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Canine Retraction
Keywords: bony changes; laser; canine retraction; CBCT

STUDY DESIGN:
Intervention Model Description: randomized double blinded clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control conventional method (Active Comparator): conventional method of canine retraction using brackets
  Interventions: Procedure: Conventional tooth movement
- study laser corticotomy (Active Comparator): an accelerated orthodontic movement using Waterlase MDTM Turbo all-tissue laser for corticotomy
  Interventions: Procedure: laser corticotomy

INTERVENTIONS:
Procedure: laser corticotomy — stimulation of tooth movement during orthodontics treatment using Waterlase MDTM Turbo all-tissue laser therapy
  Arms: study laser corticotomy
Procedure: Conventional tooth movement — tooth movement us done using wires and brackets
  Arms: control conventional method

SUMMARY:
The patient's bone morphology during orthodontic treatment is an important consideration. Therefore, during orthodontic tooth movement (OTM), an imbalance between bone resorption and deposition will cause the tooth to move out of the alveolar envelope . Unfavorable consequences like gingival recession and the dehiscence of an alveolar bone plate may arise from the movement of the teeth beyond the boundary of the bone they are housing. This happened because the dense cortical bone didn't enlarge to maintain protection for the moving root.

On the other hand, orthodontic force creates a complex loading pattern and biological response on the periodontal ligament (PDL). there was an increase in osteoclastic activity in a compression region within the PDL. In contrast, in the other tension region, there was an increase in osteoblastic activity and mineralization of the bone matrix.

DETAILED DESCRIPTION:
Orthodontic tooth movement generates complex mechanical loading patterns with corresponding complex biological responses in the periodontal tissues. This will occur only if the hard tissue around the tooth can undergo proper breakdown and build-up . The primary trigger factor responsible for orthodontic tooth movement is the strain experienced by the periodontal ligament (PDL) cells and the extracellular matrix. This strain results in alteration in the gene expression within the cells, with a production of various cytokines and chemokines, capillary vasodilatation within periodontal ligament, and migration of inflammatory cells with more cytokine production and subsequent alveolar bone remodeling in response to mechanical loading .

On application of orthodontic force, the compression region within the PDL shows increased osteoclastic activity,whereas in the tension region, there is proliferation of osteoblasts and mineralization of the extracellular matrix . In general, molecules that have been linked to tensile strains and act by stimulating osteoblast progenitor cell proliferation in the periodontal ligament, with subsequent bone formation and inhibition of bone resorption similar to orthodontic tooth movement, include transforming growth factor-beta (TGF-b), various bone morphogenic proteins (BMPs), and epidermal growth factor (EGF) . On the other hand, Interleukin-1 beta (IL-1β), interleukin-6 (IL-6), CC chemokines ligand 2 (CCL2), and other inflammatory cytokines regulate osteoclastic activity through the activation of the nuclear factor kappa B (RANK) and the nuclear factor kappa B ligand (RANKL) .

Corticotomy for rapid tooth movement was introduced in 1959 by Köle to cut the alveolar bone and move a tooth. He practiced corticotomy and osteotomy on various malocclusion cases. Vertically, the cortical and marrow bone between the teeth were partially removed, and either a subapical horizontal cut with alveolar bone cutting at a distance of one cm. from the apex or only a cortical osteotomy excluding the marrow bone was performed .

Conventional treatment with fixed appliances likely requires an average of 1.5 to 2 years, resulting in a canine retraction rate of 0.5 to 1mm per month. Therefore, other modalities have been used to accelerate OTM such as pulsed electromagnetic field, corticotomy, dento-alveolar distraction, periodontal ligament distraction, and laser therapy Laser-based technology was a dream for oral surgery to find a new tool for bone cutting. Using of pulsed erbium-doped yttrium aluminium garnet (Er:YAG) lasers showed effective cutting tool with minimum degree of carbonization. Also, it can effectively accelerate canine retraction with no complications or discomfort for the patients. The Erbium laser affects the cortical bone, leading to RAP without postsurgical complications

ELIGIBILITY:
Inclusion Criteria:

* patients who need extraction of maxillary first premolar in orthodontic treatment and patients who need canine retraction

Exclusion Criteria:

* medically compromised patient

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
assessment of labial bone thickness | 6 months
  assessment of labial bone using CBCT

SECONDARY OUTCOMES:
assessment of root length | 6 months
  assessment of root length using CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Zainab H Abdel Rahman, Phd, Principal Investigator — lecturer
Locations (1):
- Faculty of Dentistry , Al Azhar Univeristy For Girls, Cairo, Heliopolis - Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No